CLINICAL TRIAL: NCT05091970
Title: Symptom-Targeted Approach to Rehabilitation for Concussion: STAR-C
Brief Title: Symptom-Targeted Approach to Rehabilitation for Concussion
Acronym: STAR-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Texas Veterans Health Care System (U.S. Federal Agency)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); McMaster University (Other)
Responsible Party: Principal Investigator, Blessen Eapen, Chief, Physical Medicine and Rehabilitation Service, South Texas Veterans Health Care System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DoD Award: PT17006; W81XWH1820070 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2021-09-20; First posted 2021-10-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Mild Traumatic Brain Injury
Keywords: blast injuries; clinical trial; cognitive rehabilitation; concussion; mild TBI; postconcussive syndrome; posttraumatic stress disorder; traumatic brain injury
MeSH Terms: conditions — Brain Concussion; Blast Injuries; Post-Concussion Syndrome; Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-Person (Experimental): Manualized cognitive rehabilitation for mild traumatic brain injury (mTBI) delivered face-to-face.
  Interventions: Procedure: Manualized cognitive rehabilitation for mild traumatic brain injury (mTBI)
- Telehealth (Experimental): Manualized cognitive rehabilitation for mild traumatic brain injury (mTBI) delivered via telehealth.
  Interventions: Procedure: Manualized cognitive rehabilitation for mild traumatic brain injury (mTBI)

INTERVENTIONS:
Procedure: Manualized cognitive rehabilitation for mild traumatic brain injury (mTBI) — Three 60-minute sessions per week with a minimum of 6 sessions and a maximum of 10 sessions. This intervention is to be delivered by trained Occupational Therapists (OTs) and Speech-Language Pathologists (SLPs), and includes training in compensatory strategies, direct training of cognitive subskills (e.g., attention training), and assigned homework to practice skills learned in treatment.

SUMMARY:
Throughout the course of the wars in Iraq and Afghanistan, more than 250,000 service members sustained traumatic brain injuries, mostly characterized as mild traumatic brain injuries (mTBI) or concussions. While most with mTBI recover over days to weeks, a significant percentage continue to experience post-concussive symptoms such as headaches, cognitive difficulties, and dizziness for months to years. As a result, treatment of post-concussive symptoms after mTBI is of significant importance in the Department of Defense and Veterans healthcare systems.

Several studies have shown that cognitive rehabilitation can be effective for individuals with mTBI, including Service Members and Veterans with post concussive symptoms. Cognitive rehabilitation is a type of treatment in which patients work with a therapist to improve everyday memory and thinking skills and develop strategies to reduce the impact of cognitive difficulties in their everyday lives. While these treatments have great potential benefits, protocols studied to date are time intensive, requiring up to 60 hours of treatment. These time demands are impractical for many Service Members and Veterans, and place a time-burden on clinics providing the treatment.

The current study proposes to identify key ingredients of an evidence-based cognitive rehabilitation protocol to develop a streamlined version that is feasible and acceptable to Service Members and Veterans. This briefer protocol will increase the number of Service Members and Veterans who can access treatment. To accomplish this goal the investigators will first spend six months analyzing manualized treatments from a successful cognitive rehabilitation intervention developed for Service Members. The investigators will analyze manuals using a framework developed to identify active ingredients in rehabilitation. Based on those results the investigators will develop a manualized streamlined treatment protocol, which the investigators will deliver to 25 Service Members and 50 Veterans over 18 months in person or via telehealth. The investigators will determine feasibility and acceptability of this intervention, and collect preliminary efficacy data. The project addresses access to therapy services and enhanced treatment compliance, a key barrier to participation in cognitive rehabilitation by Veterans and Service Members with TBI. Additionally, although this study focuses on Service Members and Veterans with mTBI, the investigators expect that this streamlined intervention can also be translated to civilian populations with mTBI.

DETAILED DESCRIPTION:
Background

The proposed work addresses the FY17/18 PH/TBIRP CTRR-CTA Focus Area of Cognitive Rehabilitation. The study will generate new knowledge about optimal cognitive rehabilitation prescription patterns, specifically frequency (number of days), intensity (number of hours per day), and type (active ingredients). The study outcome will be a treatment protocol (STAR-C) that can be delivered efficiently and effectively in person or via telehealth, to minimize functional limitations after mTBI and maximize treatment accessibility.

The STAR-C study has features of a pragmatic trial: all individuals with mTBI are invited to enroll, regardless of co-morbidities; the primary outcome is clinically meaningful and does not require special equipment or tests; aspects of the intervention will be flexible so clinicians can tailor intervention to their clients; and there are no formal strategies to ensure compliance. Also consistent with pragmatic trial methods, the investigators will include individuals from heterogeneous practice settings (DoD and VA), and use standard-of-care outcome measures.

Mild traumatic brain injury (mTBI) is a widely acknowledged cause of morbidity among Operation Enduring Freedom and Operation Iraqi Freedom (OEF/OIF) warfighters. Several recent studies provide incidence estimates for mTBI among combat deployed troops serving in support of OEF/OIF. In a recent population cohort study, 4.9% of over 2,500 Army infantry soldiers reported mTBI with loss of consciousness, and another 10.3% reported mTBI with altered mental status. In one cross-sectional prevalence study of OEF/OIF Service Members, 12% of the sample of over 2,200 respondents to a mail survey reported a history consistent with mTBI during deployment. Recent surveillance data obtained by the Defense and Veterans Brain Injury Center (DVBIC) from electronic medical records indicate that over the past 10 years, more than 250,000 active duty Service Members have reported sustaining a TBI, with the majority of these being mild in severity.

As Service Members separate from active duty or reserve duty status, their treatment can transition to the Veterans Health Administration (VHA), which also tracks epidemiologic data. In Fiscal Year (FY) 2014, 7% of Iraq and Afghanistan War Veterans seen in the VHA system carried a diagnosis of TBI. According to Taylor et al, the prevalence of TBI diagnosis in the VA healthcare System has remained consistent since tracking began around 2009, despite changes in incidence in the DoD following the reduction of combat operations in Iraq and Afghanistan.

While mTBI is generally associated with a good prognosis for recovery, a percentage of individuals experience persistent symptoms following mTBI such as headache, dizziness and/or cognitive difficulties. The frequency of functional cognitive complaints and protracted course of symptoms are especially common in individuals with mTBI and mental health comorbidities. Regardless of the exact etiology of the symptoms, long-term cognitive complaints can impact Service Members' ability to carry out their military duties and negatively impact military readiness. Given that the central tenet of military medicine is to maintain force readiness, symptoms that affect a Service Member's ability to carry out their duties without restriction remain an important focus of treatment within the DoD Healthcare System.

For those individuals transitioning to the VA Healthcare system, effective treatment of post-concussive symptoms remains a priority. Taylor and colleagues demonstrated that VA healthcare utilization and associated costs were higher in individuals with a diagnosis of TBI compared to those without such a diagnosis (Cohen's d = .40), and although the prevalence of TBI diagnosis has remained constant, the number of individuals transitioning to the VA continues to rise. The US Department of Defense (DoD) and Veterans Health Administration (VHA) have invested significant resources in clinical treatment and treatment research for mTBI to address this important need.

There is strong evidence that cognitive rehabilitation can help reduce functional limitations for individuals with persistent cognitive symptoms after mTBI. This includes evidence from the recent DVBIC-funded Study of Cognitive Rehabilitation Effectiveness (SCORE). SCORE was a randomized controlled trial with four treatment arms: psychoeducational intervention, computer-based cognitive rehabilitation, therapist-directed cognitive rehabilitation, and a combination of therapist-directed cognitive rehabilitation plus psychotherapeutic intervention. The largest gains in functional gains were in the last two groups - i.e., when cognitive rehabilitation was delivered by a clinician, with or without psychotherapy - and benefits were maintained 3 months after treatment. SCORE was an important advance in cognitive rehabilitation for mTBI, but it had one significant limitation: the study protocol required 10 hours of individual and group therapy per week for 6 weeks. Such an extended time commitment limits the number of Service Member s and Veterans who could access treatment and increases the likelihood of patient dropout before treatment completion. As such, a shorter version of SCORE would be more practical, but until recently the investigators did not have a systematic method of identifying elements to retain or omit.

A new system for classifying rehabilitation treatments, the Rehabilitation Treatment Specification System, offers a mechanism for streamlining SCORE based on treatment principles, treatment theory, and empirical evidence. The RTSS was developed by a multidisciplinary group of rehabilitation specialists, to provide a clear and rigorous system for defining, classifying, and measuring rehabilitation treatments. The RTSS project was motivated by the lack of information about rehabilitation treatment methods, not only in research studies but also in clinical practice. While there are several systems for describing patient and study characteristics, and systems for classifying goals of treatment, these systems describe the who and what of rehabilitation. The treatments themselves, however, often are described only in terms of duration of a particular service (e.g., hours of speech therapy), or by the problems they are intended to treat (e.g., cognitive rehabilitation). What these systems do not tell us is the how of rehabilitation: what the clinician does or provides to a patient in a therapy session. The RTSS is intended to organize treatments according to these clinician actions, specifically clinician actions that are known or hypothesized to account for changes in patient functioning.

Application of the RTSS to SCORE will improve efficiency and effectiveness in three ways:

1. Ensuring a match between ingredients and targets.
2. Identifying themes across treatment activities.
3. Adding volitional ingredients.

Objectives/Specific Aims/Hypotheses:

The project aim is to use the RTSS to develop a streamlined version of the SCORE protocol (STAR-C), and then administer the STAR-C protocol to Service Members and Veterans with mTBI in person and via telehealth. The long-term goal is to improve access to cognitive rehabilitation services for Service Members, Veterans, and civilians with mTBI, to maximize return to activities and participation in meaningful life roles.

Specific objectives are:

* Objective #1: To identify core ingredients and targets in SCORE and use these to develop a Core-SCORE protocol that can be delivered 3 hours per week X 3 weeks.
* Objective #2: To complete an implementation study of STAR-C.
* Objective #3: To collect preliminary effectiveness data for a future clinical trial comparing in-person STAR-C treatment to telehealth delivery. Because access to services can be a major barrier for Service Members and Veterans, the investigators see this as a critical next step to increase access to care to Service Members and Veterans, as well as potential translation to civilian populations.

Study Design

The investigators propose an implementation study, as recommended when a previous intervention (i.e. SCORE cognitive rehabilitation trial) was successful but in a different setting than the one of interest. The SCORE results serve as pilot data for this study. The proposed study has three phases:

* Phase I (6 months): Analyze SCORE protocol using the RTSS manual to identify active ingredients and targets; and develop and manualize STAR-C protocol. Concurrently with protocol development and manualization, The investigators will complete all regulatory and Human Subjects procedures required for Phase II.
* Phase II (18 months): Implement STAR-C. Once patients are referred and pass the screening, they will be invited to participate in the study and consented using standard, approved procedures.
* Phase III (6 months): Complete collection of post-intervention implementation outcome and effectiveness data. Prepare application for a clinical trial comparing in-person to telehealth delivery of STAR-C

Target Population

The target population will be 75 adults with mTBI: 25 active duty Service Members (SMs) from the Brain Injury Rehabilitation Service at Brooke Army Medical Center (BAMC), and 50 Veterans from the San Antonio Polytrauma Rehabilitation Center at the South Texas Veterans Health Care System. mTBI will be defined according to criteria in the VA/DoD Clinical Practice Guideline for the Management of Concussion-Mild Traumatic Brain Injury and the Ohio State University TBI Identification Method (OSU TBI-ID). The treatment sample will consist of consecutive referrals to the clinic who meet inclusion criteria and consent to participate. Although our target enrollment is 75 individuals, the investigators anticipate that there will be some expected attrition. To address this issue, the investigators will recruit up to 34 SMs and 68 Veterans to ensure recruitment of the target population.

ELIGIBILITY:
Inclusion Criteria:

1. mTBI defined per the VA/DoD Clinical Practice Guideline for the Management of Concussion-Mild Traumatic Brain Injury (CPG; Corrigan & Bogner, 2007) sustained in any context (deployment-related or non-deployment-related) and at any time longer than 6 months previously;
2. A score of 3, 4, or 5 on any of the four Cognitive items on the NSI, to include participants who have cognitive complaints; and
3. A score on the Word Reading Subtest of the Wide Range Achievement Test of a sixth-grade reading level or higher, to ensure participants can read study materials.

All individuals in this study population must meet all of the inclusion criteria in order to be eligible to participate in the study

Exclusion Criteria:

1. History of TBI (any severity) within 6 months of enrollment.
2. History of a moderate, severe, or penetrating TBI as defined by DoD/VA guidelines.
3. Lifetime diagnosis of schizophrenia or other psychotic disorder.
4. Current participation in intensive behavioral health treatment (>5 appointments/encounters per week) for major depressive disorder, post-traumatic stress disorder (PTSD), bipolar disorder, or substance-related disorder.
5. History of a neurological disease other than mild TBI such as multiple sclerosis, cerebral vascular accident, brain tumor, neurodegenerative disease, or neuro-motor disorder.
6. Current, active suicidal or homicidal ideation.
7. A score of <45 on Trial 2 of the Test of Memory Malingering, or a Validity 10 score of >22 from the NSI, to exclude individuals who demonstrate suboptimal effort or potential invalid self-reporting of symptoms.
8. Daily use of narcotic pain medications.

All individuals in this study population meeting any of the exclusion criteria at baseline will be excluded from study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scaling Change | Treatment week 1, Treatment week 2, Treatment week 3, 1 week post-treatment, 4 weeks post-treatment, 12 weeks post-treatment
  Goal attainment scaling of a minimum of three goals. Score obtained for each goal at each session. Score ranges from -1 to +3. Higher numbers indicate higher levels of goal achievement.
Common Concussive Cognitive Complaints (C4) Inventory Change | Baseline; Treatment week 3 (last session); 1 week post-treatment, 4 weeks post-treatment, 12 weeks post-treatment
  23 item self-report measure that lists common post-concussive cognitive complaints. The respondent rates how often specific cognitive complaints have caused trouble for them day-to-day in the two weeks preceding the measure's administration. Item scores range from 1 = "Not at All" to 5 = "All the time"
Neurobehavioral Symptom Inventory (NSI) Change | Baseline; 1 week post-treatment, 4 weeks post-treatment, 12 weeks post-treatment
  22-item self-report checklist of persistent post-concussive symptoms and how much symptoms have disturbed the respondent since injury. Total score ranges from 0 to 88. Item response options range from 0="None" to 4 ="Very Severe"
Key Behaviors Change Inventory (KBCI) | Baseline; 1 week post-treatment, 4 weeks post-treatment, 12 weeks post-treatment
  The KBCI was designed to assess functional cognitive and behavioral changes after TBI. It is composed of 64 items rated on a 4-point scale. Response options range from "False, not at all" to "Very True"
Patient Global Impression of Change (PGIC) | Baseline; 1 week post-treatment, 4 weeks post-treatment, 12 weeks post-treatment
  Change in activity, limitations, symptoms, emotions and overall quality of life, related to painful illness. Respondents rate impression of change from 1-7, with higher scores indicating an impression of positive change, and to rate overall change on a scale ranging from 1 = "Much Better" to 10 = "Much Worse"

SECONDARY OUTCOMES:
Center for Epidemiological Studies-Depression (CES-D) | Baseline; 1 week post-treatment, 4 weeks post-treatment, 12 weeks post-treatment
  The CES-D is a 20 item self-report measure that asks respondents to rate how often in the past week they have felt symptoms related to depression on the following scale: 0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time. Positive items are reverse scored. Scores range from 0 to 60. Higher scores indicate a higher number of more frequent depressive symptoms.
Veterans Rand 36-Item Health Survey (VR-36) | Baseline; 1 week post-treatment, 4 weeks post-treatment, 12 weeks post-treatment
  36 item self-report measure that assesses level of health in domains of physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, energy/vitality, social functioning, role limitations due to emotional problems, and mental health. Higher scores indicate better ratings of health.
Epworth Sleepiness Scale - Adult Version (ESS) | Baseline; 1 week post-treatment, 4 weeks post-treatment, 12 weeks post-treatment
  The ESS is an 8-item scale that measures daytime sleepiness. Total score ranges from 0-24, with higher ratings corresponding to higher daytime sleepiness.
PTSD Checklist 5 (PCL-5) | Baseline; 1 week post-treatment, 4 weeks post-treatment, 12 weeks post-treatment
  The PTSD Checklist for DSM-5 is a 20-item self-report measure that screens for PTSD symptoms. Total score ranges from 0-80. A higher score indicates greater presence and intensity of symptoms.
Acceptability of Intervention Measure (AIM)- (Patient) | Treatment session 1(week 1), Treatment session 2 (week 1), Last Treatment session(week 3), 1 week post-treatment, 3 months post-treatment
  Acceptability ratings by patients. Scale is composed of four items rated by clinicians on a 5-point Likert scale ranging from "1 = Completely Disagree" to "5 = Completely Agree."
Acceptability of Intervention Measure (AIM)- (Clinician) | Treatment session 1(week 1), Treatment session 2 (week 1), Last Treatment session(week 3), 1 week post-treatment
  Acceptability ratings by clinicians. Scale is composed of four items rated by clinicians on a 5-point Likert scale ranging from "1 = Completely Disagree" to "5 = Completely Agree."
Intervention Appropriateness Measure (IAM) | Treatment session 1(week 1), Treatment session 2 (week 1), Last Treatment session(week 3), 1 week post-treatment
  Appropriateness ratings by clinicians. Scale is composed of four items rated by clinicians on a 5-point Likert scale ranging from "1 = Completely Disagree" to "5 = Completely Agree."
Feasibility of Intervention Measure (FIM) | Treatment session 1(week 1), Treatment session 2 (week 1), Last Treatment session(week 3), 1 week post-treatment
  Feasibility ratings by clinicians. Scale is composed of four items rated by clinicians on a 5-point Likert scale ranging from "1 = Completely Disagree" to "5 = Completely Agree."

CONTACTS AND LOCATIONS:
Overall Officials: Blessen C Eapen, MD, Principal Investigator — South Texas Veterans Health Care System; Amy O. Bowles, MD, Principal Investigator — Brooke Army Medical Center; Doug B Cooper, PhD, Principal Investigator — South Texas Veterans Health Care System
Locations (2):
- United States (2):
  - Brooke Army Medical Center, San Antonio, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belanger HG, Brown LM, Crowell TA, Vanderploeg RD, Curtiss G. The Key Behaviors Change Inventory and executive functioning in an elderly clinic sample. Clin Neuropsychol. 2002 Aug;16(3):251-7. doi: 10.1076/clin.16.3.251.13848. PMID 12607138
- [Background] Belanger HG, Lange RT, Bailie J, Iverson GL, Arrieux JP, Ivins BJ, Cole WR. [Formula: see text]Interpreting change on the neurobehavioral symptom inventory and the PTSD checklist in military personnel. Clin Neuropsychol. 2016 Oct;30(7):1063-73. doi: 10.1080/13854046.2016.1193632. Epub 2016 Jun 8. PMID 27266484
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Benge JF, Pastorek NJ, Thornton GM. Postconcussive symptoms in OEF-OIF veterans: factor structure and impact of posttraumatic stress. Rehabil Psychol. 2009 Aug;54(3):270-8. doi: 10.1037/a0016736. PMID 19702425
- [Background] Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P; CONSORT NPT Group. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 2017 Jul 4;167(1):40-47. doi: 10.7326/M17-0046. Epub 2017 Jun 20. PMID 28630973
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Center, DaVBI. DoD Worldwide Numbers for TBI. Defense and Veterans Brain Injury Center. 2017;Retrieved from http://dvbic.dcoe.mil/dod-worldwide-numbers-tbi
- [Background] Cicerone, KD., Kalmar, K. Persistent postconcussion syndrome: The structure of subjective complaints after mild traumatic brain injury. The Journal of Head Trauma Rehabilitation, 1995;10(3): 1-17.
- [Background] Cooper DB, Bowles AO, Kennedy JE, Curtiss G, French LM, Tate DF, Vanderploeg RD. Cognitive Rehabilitation for Military Service Members With Mild Traumatic Brain Injury: A Randomized Clinical Trial. J Head Trauma Rehabil. 2017 May/Jun;32(3):E1-E15. doi: 10.1097/HTR.0000000000000254. PMID 27603763
- [Background] Corrigan JD, Bogner J. Initial reliability and validity of the Ohio State University TBI Identification Method. J Head Trauma Rehabil. 2007 Nov-Dec;22(6):318-29. doi: 10.1097/01.HTR.0000300227.67748.77. PMID 18025964
- [Background] Dejong G, Horn SD, Gassaway JA, Slavin MD, Dijkers MP. Toward a taxonomy of rehabilitation interventions: Using an inductive approach to examine the "black box" of rehabilitation. Arch Phys Med Rehabil. 2004 Apr;85(4):678-86. doi: 10.1016/j.apmr.2003.06.033. PMID 15083447
- [Background] Hart T, Tsaousides T, Zanca JM, Whyte J, Packel A, Ferraro M, Dijkers MP. Toward a theory-driven classification of rehabilitation treatments. Arch Phys Med Rehabil. 2014 Jan;95(1 Suppl):S33-44.e2. doi: 10.1016/j.apmr.2013.05.032. PMID 24370323
- [Background] Helmick KM, Spells CA, Malik SZ, Davies CA, Marion DW, Hinds SR. Traumatic brain injury in the US military: epidemiology and key clinical and research programs. Brain Imaging Behav. 2015 Sep;9(3):358-66. doi: 10.1007/s11682-015-9399-z. PMID 25972118
- [Background] Hoge CW, McGurk D, Thomas JL, Cox AL, Engel CC, Castro CA. Mild traumatic brain injury in U.S. Soldiers returning from Iraq. N Engl J Med. 2008 Jan 31;358(5):453-63. doi: 10.1056/NEJMoa072972. Epub 2008 Jan 30. PMID 18234750
- [Background] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Background] Keith, RA., Lipsey, MW. The role of theory in rehabilitation assessment, treatment, and outcomes. In RL, Glueckauf, LB, Sechrest, GR, Bond, & EC, McDonel, eds., Improving Assessment in Rehabilitation and Health. Thousand Oaks, CA: Sage Publications; 1993:33-58.
- [Background] Kolitz BP, Vanderploeg RD, Curtiss G. Development of the Key Behaviors Change Inventory: a traumatic brain injury behavioral outcome assessment instrument. Arch Phys Med Rehabil. 2003 Feb;84(2):277-84. doi: 10.1053/apmr.2003.50100. PMID 12601661
- [Background] Lange RT, Brickell TA, Kennedy JE, Bailie JM, Sills C, Asmussen S, Amador R, Dilay A, Ivins B, French LM. Factors influencing postconcussion and posttraumatic stress symptom reporting following military-related concurrent polytrauma and traumatic brain injury. Arch Clin Neuropsychol. 2014 Jun;29(4):329-47. doi: 10.1093/arclin/acu013. Epub 2014 Apr 9. PMID 24723461
- [Background] Jakob R, Ustun B, Madden R, Sykes C. The WHO Family of International Classifications. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2007 Jul;50(7):924-31. doi: 10.1007/s00103-007-0281-z. PMID 17581728
- [Background] Management of Concussion/mTBI Working Group. VA/DoD Clinical Practice Guideline for Management of Concussion/Mild Traumatic Brain Injury. J Rehabil Res Dev. 2009;46(6):CP1-68. No abstract available. PMID 20108447
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Schneiderman AI, Braver ER, Kang HK. Understanding sequelae of injury mechanisms and mild traumatic brain injury incurred during the conflicts in Iraq and Afghanistan: persistent postconcussive symptoms and posttraumatic stress disorder. Am J Epidemiol. 2008 Jun 15;167(12):1446-52. doi: 10.1093/aje/kwn068. Epub 2008 Apr 17. PMID 18424429
- [Background] Soble JR, Silva MA, Vanderploeg RD, Curtiss G, Belanger HG, Donnell AJ, Scott SG. Normative Data for the Neurobehavioral Symptom Inventory (NSI) and post-concussion symptom profiles among TBI, PTSD, and nonclinical samples. Clin Neuropsychol. 2014;28(4):614-32. doi: 10.1080/13854046.2014.894576. Epub 2014 Mar 14. PMID 24625213
- [Background] Taylor, BC., Campbell, E., Nugent, S., Fletcher, L., Bidelspach, DE., Kehle- Forbes, SM., . . . Sayer, NA. Fiscal Year 2014 VA Utilization Report for Iraq and Afghanistan War Veterans Diagnosed with TBI. 2015. Retrieved from http://www.polytrauma.va.gov/TBIReports/FY14-TBI-DiagnosisHCU-Report.pdf
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. J Clin Epidemiol. 2009 May;62(5):464-75. doi: 10.1016/j.jclinepi.2008.12.011. PMID 19348971
- [Background] Turkstra LS, Norman R, Whyte J, Dijkers MP, Hart T. Knowing What We're Doing: Why Specification of Treatment Methods Is Critical for Evidence-Based Practice in Speech-Language Pathology. Am J Speech Lang Pathol. 2016 May 1;25(2):164-71. doi: 10.1044/2015_AJSLP-15-0060. PMID 27145191
- [Background] Vanderploeg RD, Belanger HG, Duchnick JD, Curtiss G. Awareness problems following moderate to severe traumatic brain injury: Prevalence, assessment methods, and injury correlates. J Rehabil Res Dev. 2007;44(7):937-50. doi: 10.1682/jrrd.2006.12.0163. PMID 18075951
- [Background] Vanderploeg RD, Silva MA, Soble JR, Curtiss G, Belanger HG, Donnell AJ, Scott SG. The structure of postconcussion symptoms on the Neurobehavioral Symptom Inventory: a comparison of alternative models. J Head Trauma Rehabil. 2015 Jan-Feb;30(1):1-11. doi: 10.1097/HTR.0000000000000009. PMID 24263177
- [Background] Warden D. Military TBI during the Iraq and Afghanistan wars. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):398-402. doi: 10.1097/00001199-200609000-00004. PMID 16983225
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Whyte J. Contributions of treatment theory and enablement theory to rehabilitation research and practice. Arch Phys Med Rehabil. 2014 Jan;95(1 Suppl):S17-23.e2. doi: 10.1016/j.apmr.2013.02.029. PMID 24370321